CLINICAL TRIAL: NCT01811875
Title: Multicentre, Non-controlled, Prospective, Post-Marketing Safety Study Following Long-Term Prophylactic OptivateTreatment in Subjects With Severe Haemophilia A
Brief Title: Post-Marketing Safety Study Following Long-Term Prophylactic OptivateTreatment in Subjects With Severe Haemophilia A
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study no longer required as Optivate German license expired in Sep-2017.
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8VWF07
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Haemophilia A
Keywords: Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — optivate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Optivate 500IU (Experimental): Optivate 500IU
  Interventions: Biological: Optivate 500IU

INTERVENTIONS:
Biological: Optivate 500IU

SUMMARY:
Primary objective: To assess post-marketing immunogenicity of Optivate® by monitoring plasma inhibitor levels for at least 100 Exposure Days (EDs) for each subject.

Secondary objectives: To assess efficacy and tolerability by monitoring FVIII recovery and adverse events

DETAILED DESCRIPTION:
The primary efficacy endpoint is to assess immunogenicity of Optivate® by monitoring plasma inhibitor level for at least 100 EDs for each subject.

FVIII inhibitor evaluation FVIII inhibitor screen data will be listed. FVIII quantitative inhibitor results will be listed. Shift tables will present the number of subjects with positive (≥ 0.6 BU) and negative (< 0.6 BU) results and those for whom the results change during the study. The number of exposure days until development of inhibitors will be summarised.

For the secondary endpoints: Descriptive statistics will be presented on the number of recoveries at each timepoint and for each subject. These will be presented for each visit and for each subject and then for each batch of FVIII/ Optivate® used. All the AE data (from CRF and study diary) will be pooled together and reported in terms of the type, duration, treatment and/or severity.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent or, if less than 18 years of age written assent (where possible) and their parent/guardian's written informed consent.
* Severe haemophilia A (< 1%# FVIII:C).
* Previously Treated Patients (PTPs) with > 150 exposure days on prior Factor VIII therapy (of which at least the last 50 EDs or 2 years treatment can be confirmed by way of subject records).
* Immunocompetent with CD4 count > 200 / µl.
* HIV negative or a viral load < 200 particles / µl.

  * subjects suffering from severe haemophilia A (<2%) may be enrolled, but only after approval by BPL. Subjects with a Factor VIII of <2% may not constitute more than 50% of the total patient population. A separate statistical evaluation will be conducted for the <1% and <2% populations.

Exclusion Criteria:

* • History of inhibitor development to FVIII or a positive result on the Nijmegen Bethesda at screening (quantitative result of > 0.6 BU) prior to the administration of Optivate®.

  * Known or suspected hypersensitivity to the investigational medicinal product or its excipients.
  * Clinically significant liver disease, renal disease, or coagulopathy other than haemophilia A.
  * History of unreliability or non cooperation (including not being able to complete the study diary).
  * Participating in, or have taken part in another trial within the last 30 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wolford, Study Director — Bio Products Laboratory
Locations (4):
- Colombia (2):
  - Fundacion BIOS, Barranquilla
  - Hospital general de Medellin, Medellín
- HZRM Haemophilia Centre Rhine Main, Darmstadt, Mörfelden-Walldorf, Germany
- Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Lodz, Poland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven patients were enrolled. One patient in Germany; 4 patients in Colombia and 2 patients in Poland.
Period: Overall Study
Arm/Group | Optivate 500IU
Started | 7
Completed | 5
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.6 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Colombia | 4
  Poland | 2
  Germany | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Did Not Develop Inhibitors to FVIII (<0.6BU)
Description: FVIII inhibitor status at any of the study visits was measured by a Nijmegen Bethesda assay and inhibitor screens. A result of ≥ 0.6 BU confirmed that the subject had developed inhibitors to FVIII. If this occurred, the test was repeated on a separate sample; if both tests were confirmed to be ≥ 0.6 BU, this was to be reported by the Investigator as a serious adverse event (SAE).
Time Frame: At least 100 Exposure Days for each subject. Subjects will attend 5 visits over a period of up to 12 months
Population: Patients who completed at least 100 exposure days to Optivate.
Measure: Count of Participants; unit: Participants
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 5
Participants | 5

2. Secondary Outcome: Recovery With Prior FVIII Concentrate (Screening Visit) Versus Recovery With First Dose With Optivate® (Visit 1) for the Protocol Population.
Description: Recovery with prior FVIII concentrate (Screening Visit) versus recovery with first dose with Optivate® (Visit 1) for the protocol population.
Time Frame: Screening and Visit 1 (up to 4 weeks)
Population: Recovery with prior FVIII concentrate (Screening Visit) versus first dose with Optivate® (Visit 1) for the protocol population.
Measure: Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 5
IU/dL per IU/kg | -0.91 [-1.87 to 0.04]

3. Secondary Outcome: Optivate® Recovery Across Visits 1 to 4 for the Protocol Population.
Description: A recovery assessment was conducted at each study visit. Recovery assessments were only conducted after a 3-day washout period and when the subject was not actively bleeding.
  At the Screening Visit, subjects who had completed a 3-day washout period and were not actively bleeding were dosed with 30 IU/kg of their prior FVIII concentrate. The dose was measured to the nearest 0.1 mL. Blood samples for the recovery assessment were to be collected at the following time points:
  * Predose
  * 15 minutes postinfusion (±5 minutes).
  * 30 minutes postinfusion (±5 minutes).
  * 1 hour postinfusion (±10 minutes). Actual times of sample collection were to be recorded in the CRF
  At visits 1, 2, 3 and 4 subjects were dosed with 30 IU/kg of Optivate and blood samples for recovery assessments were taken at the same timepoints as specified above. An ANOVA model (analysis of variance) was used to calculate the adjusted mean for recovery across visits 1 to 4.
Time Frame: Visits 1 to 4 (Up to 100 Optivate exposure days)
Measure: Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 5
IU/dL per IU/kg | -0.01 [-1.72 to 1.70]

4. Secondary Outcome: Optivate® Therapy to Treat Breakthrough Bleeds Per Subject Per Year in the Protocol Population.
Description: Optivate® therapy to treat number of breakthrough bleeds per subject per year in the protocol population over a period of 12 months.
Time Frame: Over a period of 12 months
Measure: Mean (Standard Deviation); unit: Bleeds per subject per year
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 5
Bleeds per subject per year | 3.99 (2.961)

5. Secondary Outcome: Overall Consumption of Optivate®: Number of Exposure Days for Each Subject Per Year/Subject in the Per Protocol Population.
Description: Overall consumption of Optivate®: Number of exposure days for each subject per year/subject in the per protocol population over a period of 12 months.
Time Frame: Over a period of 12 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 5
Days | 116.2 (18.12)

6. Secondary Outcome: Overall Consumption of Optivate®: Total Dose in IU/kg of Optivate® Per Subject for Prophylactic Use.
Description: Overall consumption of Optivate®: Total dose in IU/kg of Optivate® per subject for prophylactic use over a period of 12 months.
Time Frame: Over a period of 12 months
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 5
IU/kg | 3639.97 (993.464)

7. Secondary Outcome: Overall Consumption of Optivate®: Total Dose in IU/kg of Optivate® Per Subject to Treat a Bleed in the Protocol Population.
Description: Overall consumption of Optivate®: Total dose in IU/kg of Optivate® per subject to treat a bleed in the protocol population over a period of 12 months.
Time Frame: Over a period of 12 months
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 5
IU/kg | 97.72 (117.086)

8. Secondary Outcome: Overall Consumption of Optivate®: Total Number of Infusions for Prophylactic Use Per Subject in the Protocol Population.
Description: Overall consumption of Optivate®: Total number of infusions for prophylactic use per subject in the protocol population.
Time Frame: Over a period of 12 months
Measure: Mean (Standard Deviation); unit: Infusions
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 5
Infusions | 116.8 (17.66)

9. Secondary Outcome: Overall Consumption of Optivate®: Total Number of Infusions to Treat a Bleed Per Subject in the Protocol Population.
Description: Total number of infusions to treat a bleed per subject in the protocol population.
Time Frame: Over a period of 12 months
Measure: Mean (Standard Deviation); unit: Infusions
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 5
Infusions | 2.4 (3.21)

10. Secondary Outcome: Overall Consumption of Optivate®: Overall Mean Dose in IU/kg of Optivate® Per Subject/Year for Prophylactic Use in the Protocol Population.
Description: Overall consumption of Optivate®: Overall mean dose in IU/kg of Optivate® per subject/year for prophylactic use in the protocol population.
Time Frame: Over a period of 12 months
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 5
IU/kg | 3890.02 (1033.993)

11. Secondary Outcome: Treatment Emergent Adverse Events (Non-serious) in the Safety Population
Description: Treatment emergent adverse events (non-serious) in the safety population.
Time Frame: Over a period of 12 months
Population: A total of 3 patients experienced treatment emergent adverse events.
Measure: Number; unit: treatment emergent events
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 7
treatment emergent events | 5

12. Secondary Outcome: Treatment Emergent Adverse Events (Serious) in Safety Population
Description: Treatment emergent adverse events (serious) in safety population over a period of 12 months
Time Frame: Over a period of 12 months
Population: One patient experienced a treatment emergent adverse event (serious).
Measure: Number; unit: treatment emergent events
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 7
treatment emergent events | 1

13. Secondary Outcome: Number of Participants With Inhibitor Development in Safety Population (Measured by ≥0.6 Bethesda Units)
Description: Inhibitor Development: Positive FVIII inhibitor status in safety population measured by ≥0.6 Bethesda units (this was a safety measurement but was assessed as a primary efficacy endpoint).
Time Frame: Over a period of 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Optivate 500IU
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Time Frame: Over a period of 12 months
Description: Patients had an electronic diary where they could enter any adverse events they experienced in between study visits. Adverse events were assessed at each study visit otherwise. The 9 adverse events (non-serious) recorded include non-treatment emergent and treatment emergent events.
Arm/Group | Optivate 500IU
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optivate 500IU (N=7)
Fatal road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optivate 500IU (N=7)
COMMON COLD (Infections and infestations) | 1 (1)
ANKLE TRAUMA (Injury, poisoning and procedural complications) | 1 (1)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SOFT TISSUE TRAUMA LEFT HAND (Injury, poisoning and procedural complications) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
HEMARTHROSIS OF RIGHT ELBOW (Musculoskeletal and connective tissue disorders) | 1 (1)
GENERAL PAIN (General disorders) | 1 (1)
JOINT PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
HEMARTHROSIS OF RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-11-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT01811875/Prot_000.pdf
  • Statistical Analysis Plan (2013-05-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT01811875/SAP_001.pdf